CLINICAL TRIAL: NCT03194906
Title: Memantine for Prevention of Cognitive Late Effects in Pediatric Patients Receiving Cranial Radiation Therapy for Localized Brain Tumors: A Pilot Study
Brief Title: Memantine for Prevention of Cognitive Late Effects in Pediatric Patients Receiving Cranial Radiation Therapy for Localized Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MEMCRT; R21CA218625 (NIH); NCI-2017-01279 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Glioma of Brain; Craniopharyngioma; Ependymoma; Germ Cell Tumor
Keywords: Pediatric oncology; Brain tumor; Low grade glioma; Cognitive late effects; Radiation therapy; Neuroprotection; Memantine
MeSH Terms: conditions — Craniopharyngioma; Ependymoma; Neoplasms, Germ Cell and Embryonal; Brain Neoplasms | interventions — Memantine; Medication Errors; Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Memantine (Active Comparator): Beginning at least two weeks prior to radiation therapy, participants receive memantine. Treatment continues for 12 weeks with periodic cognitive assessments and lab work.
  Interventions: Drug: Memantine; Other: Cognitive Assessment
- Placebo (Placebo Comparator): Beginning at least two weeks prior to radiation therapy, participants receive a placebo. Treatment and assessment are identical to the memantine group.
  Interventions: Other: Placebo; Other: Cognitive Assessment

INTERVENTIONS:
Drug: Memantine — Medication dosing will be overseen by one of the study neurologists, with step-wise dose reductions (5 mg intervals) allowable in the case of side effects.
  Other Names: Memantine hydrochloride; Namenda®
  Arms: Memantine
Other: Placebo — A placebo that appears exactly like the study drug, memantine, will be given in a manner identical to the study drug.
  Other Names: Look-alike drug
  Arms: Placebo
Other: Cognitive Assessment — Cognitive and neurologic examinations will be conducted to assess cognitive, social, quality of life, and neurological outcomes associated with memantine will be completed at baseline prior to medication start, and at 6 weeks (end of radiation therapy), 12 weeks (discontinuation of study medication or placebo), and one year post radiation therapy.
  Other Names: Cognitive and neurologic examinations

SUMMARY:
Children with brain tumors who have had radiation therapy are at risk for problems with attention, memory, and problem solving. Such problems may cause difficulty in school and daily life. Memantine, the drug being used for this study, is not yet approved for use in children by the U.S. Food and Drug Administration. However, studies have shown some improvements in memory for patients with dementia, Attention Deficit Hyperactivity Disorder, and autism. Scientists have also used this medication for adult cancer patients receiving radiation therapy with results showing less cognitive declines over time compared to patients taking a placebo (inactive pill). These studies have also shown few side effects.

This is a pilot/feasibility study and the first known study involving children with a cancer diagnosis or brain tumor.

PRIMARY OBJECTIVES:

* To estimate the participation rate in a study of memantine used as a neuro-protective agent in children undergoing radiotherapy for localized brain tumors (low grade glioma, craniopharyngioma, ependymoma, or germ cell tumor)
* To estimate the rate of memantine medication adherence
* To estimate the rate of completion of cognitive assessments

SECONDARY OBJECTIVES:

* To estimate the effect size of change in neurobehavioral outcomes (cognitive, social, quality of life, neurologic) associated with memantine
* To evaluate the frequency and nature of memantine side effects as measured by the Systematic Assessment for Treatment Emergent Events (SAFTEE)

DETAILED DESCRIPTION:
Participants will be randomized to take part in one of two groups:

* The Memantine Group will be prescribed memantine at a dosage following FDA-approved adult labeling. A low dose will initially be given beginning at least two weeks (± 7 days) prior to beginning radiation therapy. The dose will increase until participants reach the target dose of 20 mg/day. Memantine will be given for a total of 12 weeks.
* The Placebo Group will be prescribed identical capsules with no active drug. The placebo drug will be given in the same dose and frequency as described for the Memantine group.

Participants will undergo the same evaluations and monitoring throughout the medication phase. Assessments will be done at baseline prior to study start, with follow-up assessments at 6 weeks (end of radiation therapy), and 12 weeks (end of study medication). Psychological testing to measure attention, working memory, problem solving, intelligence and academics will be done for each participant. Caregivers will also complete questionnaires about attention, problem solving, mood and interpersonal interactions. Caregivers will also be asked to complete a questionnaire about the family's general characteristics and medical history.

At the time points noted above, blood work, vital signs and echocardiograms will be obtained, and the study neurologist will examine the participant to monitor side effects and neurological functioning. A study nurse will contact the participant once per week during the 12 weeks of medication administration to identify possible medication-related side effects and to check on rate of compliance with taking the medication. A remote app will be installed on the participant's home computer or cell phone to help remind them to take the medication and track success. At one year post medication, psychological and neurological examinations will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to 21 years at time of study enrollment
* Diagnosis of localized low grade glioma [e.g., pilocytic astrocytoma, optic pathway glioma, ogligodendroglioma, ganglioglioma, pleomorphic xanthoastrocytoma (PXA)], craniopharyngioma, ependymoma, or germ cell tumor
* Initiating focal cranial radiation therapy (photon or proton)
* Laboratory tests [transaminases (ALT, AST, ALP), BUN and creatinine not greater than twice normal] and normal ECG
* Speak, read and understand English sufficiently to complete study assessments
* Adequate vision and hearing for valid completion of study measures
* Negative βHCG pregnancy test among females of childbearing age
* Participant must be able to swallow pills (psychology staff will be available to assist with pill swallowing training if needed)
* Parent/Legal guardian available and able to speak, read and understand English

Exclusion Criteria:

* Medical disorder that would endanger subject's well-being (e.g., uncorrected hypothyroidism, cardiac arrhythmia, hypertension requiring treatment, sick sinus syndrome, prolonged QTc)
* History of significant neurological disease including poorly controlled seizures (i.e., > 1 seizure per month; anti-epileptic medications are acceptable), stroke, or head injury with loss of consciousness
* Psychiatric condition that would preclude or take precedence over study participation (e.g., active psychosis, suicidal ideation)
* IQ below 70 based on baseline/screening assessment
* Treatment with psychotropic medication (psychostimulant, antidepressant, anxiolytic, antipsychotic) within the past two weeks, unless being prescribed specifically as an anti-emetic
* History of substance abuse
* History of hypersensitivity or reaction to NMDA receptor antagonists
* History of prior cranial radiation therapy

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Percent of approached participants who consent to study participation | Once, prior to enrollment
  The rates of study participation and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 60%. The rate will be evaluated for the group as a whole as well as separately for the memantine intervention and placebo-control groups.
Percent of participants who complete all 12 weeks of memantine/placebo therapy | At completion of memantine/placebo therapy (12 weeks)
  The rates of medication adherence and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 80%. The rate will be evaluated for the group as a whole as well as separately for the memantine intervention and placebo-control groups.
Percent of participants who complete at least 3 of 4 cognitive assessments | At end of study (up to one year after study enrollment)
  The rates of completion of cognitive assessments and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 75%. The rate will be evaluated for the group as a whole as well as separately for the memantine intervention and placebo-control groups.

SECONDARY OUTCOMES:
Change in neurobehavioral outcome | At baseline (prior to start of therapy) compared at end of radiation therapy (6 weeks later)
  The effect size (Cohen's d- the standardized difference between two means) of memantine on neurobehavioral outcomes (cognitive, social, quality of life, neurologic) will be estimated by comparing performance at baseline to performance at 6 weeks (end of radiation therapy) using paired difference divided by its estimated standard deviation. In addition, due to the missing data, mixed-effects models will be fitted to investigate the change of outcome from baseline to 6 weeks.
Change in neurobehavioral outcome | At baseline (prior to start of therapy) compared at end of medication trial (12 weeks later)
  The effect size (Cohen's d- the standardized difference between two means) of memantine on neurobehavioral outcomes (cognitive, social, quality of life, neurologic) will be estimated by comparing performance at baseline to performance at 12 weeks (end of medication trial) using paired difference divided by its estimated standard deviation. In addition, due to the missing data, mixed-effects models will be fitted to investigate the change of outcome from baseline to 12 weeks.
Change in neurobehavioral outcome | At baseline (prior to start of therapy) compared at follow-up (up to 1 year later)
  The effect size (Cohen's d- the standardized difference between two means) of memantine on neurobehavioral outcomes (cognitive, social, quality of life, neurologic) will be estimated by comparing performance at baseline to performance at follow-up (up to 1 year) using paired difference divided by its estimated standard deviation. In addition, due to the missing data, mixed-effects models will be fitted to investigate the change of outcome from baseline to 1 year.
Frequency of memantine side effects | From start of memantine/placebo therapy through end of therapy (up to 12 weeks later)
  The frequency and nature of memantine side effects as measured by the SAFTEE will be evaluated qualitatively by calculating the frequency of side effect reporting by severity rating at different time points in the medication trial and comparing these frequencies across the memantine intervention and placebo-control groups. The frequency of side effects will be compared between the intervention and placebo-control groups using at t-test or other appropriate test, depending on the data distribution features of the compared outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M. Conklin, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols